CLINICAL TRIAL: NCT04831203
Title: An Egg-protein Hydrolysate (NWT-03) to Boost Brain Function - Mind Your Blood Vessels
Brief Title: NWT-03 and Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC 20-092
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-08

CONDITIONS: Brain Vascular Function; Cognition
Keywords: Cerebral Blood Flow; Cognitive Performance
MeSH Terms: interventions — NWT-03

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-hydrolysate (Experimental): Dietary supplement: an egg-protein hydrolysate (NWT-03) Study volunteers will receive a daily powder of 5 g of protein hydrolysate to mix with 200 mL of water for 36 weeks.
  Interventions: Dietary Supplement: An egg-protein hydrolysate (NWT-03)
- Control (Placebo Comparator): Control: 5 g of maltodextrin powder mixed with 250 mL of water for 36 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: An egg-protein hydrolysate (NWT-03) — As described in the experimental arm
  Arms: Protein-hydrolysate
Dietary Supplement: Placebo — As described in the Control arm
  Arms: Control

SUMMARY:
Age-related chronic diseases including dementia, type II diabetes mellitus (T2DM) and cardiovascular disease (CVD) become more prevalent and of increasing societal concern. Common denominators of these co-morbidities are insulin-resistance and impaired vascular function. Animal and short-term human studies now suggest that NWT-03 - an egg-protein hydrolysate - improves insulin-sensitivity and peripheral vascular function, which are risk markers for the development of T2DM and CVD. Insulin-resistance is also associated with cognitive decline, while impaired brain vascular function is an important event preceding the development of impaired cognitive performance. The investigators have already shown in a shorter-term trial (12 weeks) beneficial effects of a daily dose of 5.0 g of NWT-03 on cognitive performance. However, underlying mechanisms have not yet been addressed, while the long-term effects remain unknown. Thus, the investigators now hypothesize that NWT-03 beneficially affects cognitive performance and brain vascular function following long-term daily intake.

The primary objectives of this trial are to evaluate in overweight or obese adults (aged 60-75) with subjective cognitive decline (SCD) the effects of a 36-weeks NWT-03 intervention on (1) cognitive performance using a neurophysiological test battery, and (2) cerebral blood flow, as quantified by the current non-invasive gold standard magnetic resonance imaging (MRI) perfusion method Arterial Spin Labeling (ASL). Secondary study objectives are to examine effects on insulin-sensitivity and peripheral vascular function.

This intervention study will have a randomized, controlled, parallel design. The total study duration will be 36 weeks. Forty-four older adults (aged 60-75 years) with a Body Mass Index (BMI) between 25-35 kg/m2 (overweight or obese) and subjective cognitive decline (SCD), as assessed with the cognitive failure questionnaire, will participate. These study individuals are known to be at increased risk of cognitive impairment, allowing for improvement by the intervention. During the study, subjects will receive daily (in the morning) 5.0 g NWT-03 or placebo powders for 36 weeks.

DETAILED DESCRIPTION:
Due to the aging population, the number of people with cognitive impairment will have doubled by the year 2035. Also, the number of individuals with type-2 diabetes mellitus (T2DM) and cardiovascular disease (CVD) will have increased substantially. Common denominators of these age-related co-morbidities in humans are insulin-resistance and an impaired vascular function.

Newtricious (NWT)-03 is a novel dietary egg-protein hydrolysate that has proven benefits on glucose and insulin metabolism, as the investigators have recently shown in overweight or obese individuals with T2DM or impaired glucose tolerance. Furthermore, peripheral vascular function was improved. The potential explanation of these effects may arise from the finding that NWT-03 blocks the enzyme dipeptidyl peptidase (DPP)-IV (7) - a pharmaceutical target for the treatment of T2DM and CVD - that beneficially affects insulin metabolism. Compared to the wealth of knowledge about the impact of insulin-sensitivity and peripheral vascular function on the risk of T2DM and CVD, emerging evidence also indicates that these risk markers affect cognitive performance. This is of great interest, since the brain is an insulin sensitive organ and insulin-resistance is associated with cognitive decline, while impaired brain vascular function is a key pathophysiological event preceding the development of an impaired cognitive performance. A study in mice also showed effects of NWT-03 on neuro-inflammation and oxidative stress in the brain. In fact, a decreased expression of TNF-α and improved expression of enzymes involved in anti-oxidative processes were observed. The investigators have also shown in a similar - but shorter-term (12 weeks) - trial beneficial effects of NWT-03 on executive function, as the latency of response was reduced (manuscripts in preparation). In addition, the hen egg-white hydrolysate (i.e. LumiVida) also improved reaction time in middle-aged women. Underlying mechanisms of these hydrolysates on cognitive performance were however not addressed. In our review the investigators summarized the impact of dietary factors and exercise on brain vascular function in adults and discussed the relation between these effects with changes in cognitive performance. It was concluded that studies on the longer-term effects of lifestyle factors, including diet and physical exercise, can improve brain vascular function, which may contribute to the beneficial effects observed on cognitive performance. In addition, longer-term effects remain unknown and only a limited number of parameters related to cognitive performance were studied. Therefore, the investigators propose to perform a long-term placebo-controlled double blind intervention study including functional outcome parameters and study in vivo effects of NWT-03 on brain vascular function, which is a potential target to prevent or slow-down cognitive impairments, and improve cognitive performance. Focus will be on older adults (aged 60-75 years) with a Body Mass Index (BMI) between 25-35 kg/m2 (overweight or obese) and subjective cognitive decline (SCD), as assessed with the cognitive failure questionnaire. These individuals are known to be at increased risk of cognitive impairment, allowing for improvement by the intervention.

Secondary study endpoints are effects on insulin-sensitivity and peripheral vascular function, which are risk markers that may affect cognitive performance. Finally, the investigators will focus on other potential mechanisms underlying effects on brain function (i.e. ambulatory blood pressure, structural brain status, humoral factors, and the more conventional cardiometabolic risk markers) and other perceivable benefits, including general well-being (quality of life, sleep characteristics and mood) and physical fitness.

Effects will be investigated using innovative and emerging non-invasive brain magnetic resonance imaging (MRI)-perfusion methods, while focusing on whole brain and cognitive-control brain areas plus cognitive performance tests. Furthermore, the investigators have reviewed that cerebral blood flow in gray matter is a sensitive and straightforward marker of brain vascular function, which correlates with cognitive performance. Of note, lower cerebral blood flow is associated with accelerated cognitive decline and increased risk of dementia in the general population based on results of the Rotterdam prospective cohort study. Cerebral blood flow changes will be quantified on a Siemens 3 Tesla Magnetom Prisma Fit scanner at the Scannexus research facilities by the non-invasive gold standard approach: the MRI perfusion method pseudo-continuous Arterial Spin Labeling.Cognitive performance will be assessed using CANTAB (i.e. Cambridge Neuropsychological Test Automated Battery). These validated assessments for state-of-the-art cognitive testing focus on the main cognitive domains (i.e. executive function, attention and memory). Brain vascular function will be investigated using innovative and emerging non-invasive brain magnetic resonance imaging (MRI)-perfusion methods, while focusing on whole brain and cognitive-control brain areas plus cognitive performance tests. Furthermore, the investigators have reviewed that cerebral blood flow in gray matter is a sensitive and straightforward marker of brain vascular function, which correlates with cognitive performance. Of note, lower cerebral blood flow is associated with accelerated cognitive decline and increased risk of dementia in the general population based on results of the Rotterdam prospective cohort study. Cerebral blood flow changes will be quantified on a Siemens 3 Tesla Magnetom Prisma Fit scanner at the Scannexus research facilities by the non-invasive gold standard approach: the MRI perfusion method pseudo-continuous Arterial Spin Labeling.

Considering the background information given in the previous paragraph, the following research questions are formulated:

Primary research question:

What are the effects in older adults with a BMI between 25-35 kg/m2 and SCD of a 36-weeks NWT-03 intervention on (i) cognitive performance using a neurophysiological test battery, and (ii) cerebral blood flow, as quantified by the MRI-perfusion method Arterial Spin Labelling?

Major null hypotheses, H0:

1. A 36-weeks NWT-03 intervention does not significantly affect cognitive performance in older adults with a BMI between 25-35 kg/m2 and SCD.
2. A 36-weeks NWT-03 intervention does not significantly affect cerebral blood flow, as assessed by Arterial Spin Labelling, in older adults with a BMI between 25-35 kg/m2 and SCD.

Major alternate hypotheses, Ha:

1. A 36-weeks NWT-03 intervention significantly affects cognitive performance in older adults with a BMI between 25-35 kg/m2 and SCD.
2. A 36-weeks NWT-03 intervention significantly affects cerebral blood flow, as assessed by Arterial Spin Labelling, in older adults with a BMI between 25-35 kg/m2 and SCD.

Secondary research question:

What are the effects in older adults with SCD of a 36-weeks NWT-03 intervention on insulin sensitivity and peripheral vascular function, which are risk markers for T2DM and CVD?

Exploratory research questions:

What are the effects in older adults with subjective cognitive decline (SCD) of a 36-weeks NWT-03 intervention on;

* mechanisms underlying effects on brain function, including structural brain status, humoral factors, and the more conventional cardiometabolic risk markers;
* perceivable (consumer) benefits, including physical fitness and general well-being.

A randomized, placebo-controlled trial with a parallel design will be conducted.

Before screening, subjects will be informed about the procedures and informed consent will be obtained. Following screening, study participants that fulfill all inclusion criteria and are willing to participate will be asked to participate in this study.

Subjects will be informed about their screening results, including anthropometric measures (weight, length, body mass index), systolic and diastolic blood pressure (SBP and DBP), serum total cholesterol and triacylglycerol concentrations, and plasma glucose concentrations. When treatment with drugs or lifestyle interventions is indicated according to the Standards of the Dutch general practitioners' community (NHG), subjects will be advised to consult their general practitioner. Study results obtained during the intervention trial (i.e. brain vascular function) will be reported in a descriptive way at a group level, for example: "brain vascular function is improved". because no accepted normal ranges exist for these measurements.

On the days before blood sampling, adults are asked not to perform any strenuous physical exercise or to consume alcoholic beverages. On the morning of blood sampling - after a 12-hour overnight fast (from 8.00 PM) - study subjects are only allowed to drink a glass of water. Subjects are also asked not to change their habitual diet during the study. Finally, subjects are asked to come to the Metabolic Research Unit (MRUM) by public transport or car (and not by foot or bike) to standardize research measurements as much as possible

At baseline and after 18 weeks, anthropometric measurements will be performed, and a fasting blood sample will be drawn. At baseline and after 36 weeks, subjects have to attend two times the research facilities to perform the follow-up measurements: once for the "Day A" measurements and once for the "Day B" measurements. During these tests, study participants have to stay at the university and are not allowed to eat. These test days will take place with an interval of three days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 60-75 years
* Subjective cognitive decline (SCD)
* BMI between 25-35 kg/m2
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L (further testing will be performed for excessive hyperlipidemia [serum total cholesterol ≥ 8.0 mmol/L] according to the Standard for cardiovascular risk management of NHG)
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Left-handedness
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic units per day
* Use of vitamin or mineral supplements known to interfere with the main outcomes as judged by the principal investigators within the previous 1-month
* Use of medication to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g. pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Brain Vascular Function | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)
Cognitive performance | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Cambridge Neuropsychological Test Automated Battery (CANTAB)

SECONDARY OUTCOMES:
Glucose metabolism | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Oral Glucose Tolerance Test (OGTT)
Peripheral vascular function (1) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Flow-mediated vasodilation (FMD)
Peripheral vascular function (2) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Carotid artery reactivity (CAR)
Peripheral vascular function (3) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Pulse wave analysis (PWA)
Peripheral vascular function (4) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Pulse wave velocity (PWV)
Peripheral vascular function (5) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Retinal microvascular calibers

OTHER OUTCOMES:
Systolic and Diastolic Blood pressure | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Office and 24-hour ambulatory blood pressure
Advanced glycation endproducts | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Serum protein-bound advanced glycation endproducts (AGEs)
Blood lipids | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Lipids and Lipoproteins
Blood glucose | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Glucose
Blood Insulin | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  insulin
Blood markers for low-grade systemic inflammation | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Markers for low-grade systemic inflammation (IL-6, TNF-alpha)
Blood markers for microvascular function | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Markers for microvascular function (sCAM-1, vWf, cGMP)
Blood marker of neurogenesis | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Brain-derived neurotrophic factor
Structural brain status | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  MRI Structural MPRAGE scan
Other perceivable benefits: Quality of Life | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  The Quality of life will be assessed using a 32-item questionnaire
Other perceivable benefits: Physical fitness (1) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Timed up-and-go test (TUGT)
Other perceivable benefits: Physical fitness (2) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  The 6-minute walk test (6 MWT)
Other perceivable benefits: Physical fitness (4) | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Muscle strength test, as measured using the Biodex system
Weight | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Weight in kg
Height | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Height in kg
Waist circumference | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Waist circumference in centimeters
Hip circumference | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Hip circumference in centimeters
Indirect fat distribution | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Measured by skinfold measurements
Food intake | Change in outcomes at the end of a 36-week protein hydrolysate intervention and 36-week control period
  Food intake will be assessed using the Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Adams MS, Mensink RP, Plat J, Winkens B, Joris PJ. Long-term egg-protein hydrolysate consumption improves endothelial function: a randomized, double-blind, placebo-controlled trial in older adults with overweight or obesity. Eur J Nutr. 2024 Dec 24;64(1):54. doi: 10.1007/s00394-024-03566-w. PMID 39718599